CLINICAL TRIAL: NCT02767362
Title: Evaluating the Anti-Proliferative Effects of Atorvastatin on the Endometrium of Endometrial Cancer Patients: A Pre-Operative Window Study
Brief Title: A Pre-Op Window Study Evaluating Anti-Proliferative Effects of Atorvastatin on the Endometrium
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Wilma Williams Education and Clinical Research for Endometrial Cancer Award (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1514
Record Dates: First submitted 2015-11-23; First posted 2016-05-10 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Endometrial Cancer
Keywords: atorvastatin; endometrium; endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Atorvastatin; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Patients will undergo atorvastatin treatment for a minimum of 2 weeks but no more than a maximum of 4 weeks prior to surgery. At the time of hysterectomy and surgical staging, women will undergo repeat endometrial biopsy in the operating room under general anesthesia.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Once enrolled on this pre-operative window study, patients with endometrial cancer will be treated with the standard clinical dose of atorvastatin (80 mg once daily orally) for an average of 2-4 weeks prior to surgical staging. Patients will need to be able to undergo atorvastatin treatment for a minimum of 2 weeks but no more than a maximum of 4 weeks prior to surgical staging.
  Other Names: Ezetimibe

SUMMARY:
This is a preoperative window, phase 0 study of short-term atorvastatin treatment in obese women who are to undergo surgical staging for endometrial cancer.

DETAILED DESCRIPTION:
This is a preoperative window, phase 0 study of short-term atorvastatin treatment in obese women who are to undergo surgical staging for endometrial cancer. After recruitment is completed, 24 paired endometrial biopsies and hysterectomy specimens from endometrial cancer patients treated at University of North Carolina at Chapel Hill will be retrospectively obtained from the Department of Pathology to serve as controls. These cases will be matched for stage and grade to the endometrial cancers of those women enrolled on this phase 0 clinical trial and will undergo the same immunohistochemical analysis. Two previous phase 0 window studies of metformin in endometrial cancer have found no difference in Ki-67 expression between preoperative endometrial biopsy and hysterectomy specimen in control patients, although a difference was seen in metformin treated patients. However, the investigators plan to include a control group to ensure that changes found between pre- and post-atorvastatin treated patients are due to the effects of this drug versus differences in the type of specimen examined (i.e. endometrial biopsy specimen obtained in clinic versus hysterectomy specimen obtained at the time of surgery). In addition, enrolled patients will undergo repeat endometrial biopsy post- atorvastatin treatment at the time of their surgical staging. Thus, study investigators plan to compare pre-treatment endometrial biopsies to both post-treatment endometrial biopsies and hysterectomy specimens as well as have a historical control group.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-75 years old
* Have a confirmed diagnosis of type I endometrial cancer (endometrioid) based on pre-operative endometrial biopsy or dilation and curettage (D&C)
* Have a BMI >30
* Have no contraindication to short-term atorvastatin therapy
* Have a serum creatinine ≤ 1.0 mg/dL
* Have normal serum transaminase values (AST and ALT)
* Need to be able to undergo atorvastatin treatment for a minimum of 2 weeks but no more than a maximum of 4 weeks prior to surgical staging

Exclusion Criteria:

* Are currently taking a statin or have taken a statin in the past 6 months or have a history of an allergic reaction or intolerance at any time to a statin
* Have a history of liver or renal dysfunction
* Have a history of alcoholism
* Are pregnant
* Are currently taking any hormonal therapy or have been on hormonal therapy in the past 4 weeks
* Are taking a drug that may significantly interact or influence the metabolism of atorvastatin
* Concomitant cyclosporine, gemfibrozil, telaprevir, or tipranavir/ritonavir use
* History of stroke or transient ischemic attack in the preceding 6 months

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11; Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Absolute difference score | Two Years
  Measurement of the change in tumor proliferation as measured by Ki67 immunohistochemical staining after 2-4 weeks of treatment with atorvastatin. For visual comparisons of pre- and post-treatment measures, informative plots will be generated. For statistical comparisons of pre- and post-treatment measures absolute difference scores will be created. An absolute difference score is the subtraction of a post-treatment measurement from a pre-treatment measurement. The nonparametric Wilcoxon signed-rank tests will be used to examine the significance of the absolute difference scores for each measure of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Clark, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina at Chapel Hill Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org